CLINICAL TRIAL: NCT06993051
Title: Social-HEROES: Health and Education on Research Opportunities Empower Students and Tackle Inequalities
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Helena Rafaela Vieira do Rosario, PhD, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U. Minho; LCF/PR/SR24/57010020 (Other Grant/Funding Number: "la Caixa" Foudation)
Record Dates: First submitted 2025-05-07; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Overweight; Obesity
Keywords: Health Promotion, Health Literacy, Life Style, Diet, Motor Activity, Sedentary Behavior, Sleep, Child Development, Health Equity, Noncommunicable Disease
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Sedentary Behavior; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Cluster-randomized (preschool-level) parallel assignment with two arms (intervention vs. control).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Education Control (No Intervention): Preschools (n = 5; ~ 239 children) continue their usual curriculum and health-education practices; no additional components are delivered.
  No intervention will occur.
- Social-HEROES Intervention (Experimental): Six-month, cluster-level programme co-created in participatory innovation labs. Includes classroom activities and family workshops to improve diet, 24-h movement (physical activity, sedentary time, sleep) and socio-emotional skills. Implemented in 5 preschools (~ 239 children).
  Interventions: Behavioral: Social-HEROES Health-Promotion Program

INTERVENTIONS:
Behavioral: Social-HEROES Health-Promotion Program — Six-month, cluster-level, stakeholder-co-created health-promotion programme delivered in preschool settings. The programme is developed through participatory innovation labs and includes:
  * Educator training sessions (monthly)
  * Classroom activities on healthy eating, active play and socio-emotional skills (weekly)
  * Family workshops and take-home materials promoting 24-hour movement behaviour (diet, physical activity, reduced sedentary time, adequate sleep) (every 4-6 weeks)
  * Community engagement events (beginning and end of intervention). Implementation period: 6 months; dosage approx. 20-24 contact hours per child.
  Arms: Social-HEROES Intervention

SUMMARY:
Social-HEROES (Social Health and Education Research Opportunities: Empower Students and tackle inequities) is a cluster-randomised study that aims to improve the health of vulnerable preschool children (3 to 6 years old) attending Portuguese TEIP* schools.

Ten preschools (about 478 children) will be randomly assigned to one of two groups. Five preschools (≈ 239 children) will continue with their usual educational activities (control group). The other five preschools (≈ 239 children) will take part in a six-month "Social-HEROES" programme (intervention group).

The intervention is created in participatory innovation labs where children, educators, families, community members and policy-makers design activities together, guided by a systems-thinking approach. These activities encourage healthier eating, more balanced 24-hour movement (active play, less sitting, better sleep) and stronger socio-emotional skills.

The study pursues two main goals. First, it will develop this innovative, stakeholder-driven health-promotion programme. Second, it will test how well the programme works by measuring: (a) children's health-literacy levels, (b) their lifestyle habits (diet, physical activity, sedentary time and sleep), (c) rates of overweight and obesity, and (d) blood-pressure levels.

Researchers expect that, compared with the control group, children in the intervention group will show higher health-literacy scores, healthier lifestyle patterns and lower rates of excess weight and raised blood pressure. Data will be collected before the programme starts and again six months later, using short questionnaires, simple body measurements, blood-pressure readings and a wrist-worn activity tracker (accelerometer) worn for seven days. Participation is voluntary, can be stopped at any time without penalty, and all information is handled in accordance with GDPR.

Social-HEROES is funded by Fundación "la Caixa" (LCF/PR/SR24/57010020) and has ethical approval from the Life and Health Sciences Research Ethics Committee (CEICVS 189/2024). It addresses two pressing challenges at once: reducing early non-communicable-disease risks and narrowing social and educational health gaps among young children.

*TEIP: Priority Intervention Educational Territories in Portugal

ELIGIBILITY:
Inclusion Criteria:

* Children from TEIP schools
* Ages between 3 to 6 years old

Exclusion Criteria:

* Children/families who don't speak/understand Portuguese

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 478 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overweight and obesity | 6 months
  Weight (kg) and height (m) will be measured by trained staff and used to calculate body mass index (BMI = kg/m²). Values will be converted into BMI-for-age z-scores using the WHO 2006 growth standards.
Risk of high blood pressure | 6 months
  Blood pressure percentile - Systolic and diastolic blood pressure will be measured using a validated paediatric oscillometric device. Percentiles adjusted for age, sex and height will be calculated according to AAP 2017 guidelines.
Health literacy | 6 months
  Assessed using the Health Literacy Survey for Children (HLS-Child), a 20-item scale scored from 1 (very difficult) to 4 (very easy). Total score range: 20 to 80. Higher scores indicate better health literacy.

SECONDARY OUTCOMES:
Dietary intake - fruit and vegetables | 6 months
  Mean daily servings of fruits and vegetables will be estimated through a parent-completed 24-hour dietary recall. Unit: servings/day.
Dietary intake - sugar-sweetened beverages | 6 months
  Daily consumption of sugar-sweetened beverages will be estimated through a parent-completed 24-hour dietary recall. Unit: millilitres/day.
Physical activity | 6 months
  Moderate-to-vigorous physical activity (MVPA) Assessed using wrist-worn ActiGraph GT3X+ accelerometers over 7 consecutive days. Activity counts per minute will be processed using validated cut-points to calculate average daily MVPA. Unit: minutes/day.
Sedentary time | 6 months
  Accelerometer data from the same 7-day period will be analysed to estimate sedentary behaviour, defined as <100 counts per minute. Unit: minutes/day.
Sleep duration | 6 months
  Nightly sleep duration will be estimated using the Sadeh algorithm applied to 7-day ActiGraph GT3X+ wrist accelerometer data. Unit: hours/night.
Sleep quality | 6 months
  Assessed using the Portuguese version of the Children's Sleep Habits Questionnaire (CSHQ-PT), which includes 33 items scored from 1 (rarely) to 3 (usually). Total score range: 33 to 99. Higher scores indicate poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minho, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No